CLINICAL TRIAL: NCT01500915
Title: FUSION Regimen: A Disease Activity Guided Treatment Algorithm With Ranibizumab in naïve Subjects With Exudative Age-related Macular Degeneration
Brief Title: FUSION Regimen: Combined Pro re Nata and Fixed Regimen Ranibizumab in Exudative Age-related Macular Degeneration
Acronym: FUSION
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Institut de la Macula y la Retina (Other)
Collaborators: Centro Medico Teknon (Other)
Responsible Party: Principal Investigator, Jordi Mones, Director, Institut de la Macula y la Retina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FUSION-001-10-2010
Record Dates: First submitted 2011-12-14; First posted 2011-12-29 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Exudative Age-related Macular Degeneration
Keywords: AMD; ranibizumab; antiVEGF; regimen of injections; anti VEGF regimen; PRN; treat and extend
MeSH Terms: interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ranibizumab (Experimental)
  Interventions: Drug: Ranibizumab

INTERVENTIONS:
Drug: Ranibizumab — 0,5mg intravitreal ranibizumab
  Other Names: luncentis

SUMMARY:
The purpose of this study is to investigate the safety and efficacy of a combined fixed-interval and a pro re nata (PRN) regimens of ranibizumab (FUSION regimen) for the treatment of exudative age-related macular degeneration (AMD) in patients with good visual acuity (VA) at baseline. To establish whether similar efficacy to monthly regimens can be achieved with fewer injections, even in patients with good VA.

DETAILED DESCRIPTION:
This is a prospective, open-label, consecutive interventional case series in treatment-naïve patients with exudative AMD. A loading phase of 2-3 injections is followed by a fixed-interval regimen of injections combined with a pro re nata regimen for 12 months. Endpoints include VA, presence of fluid at spectral domain optical coherent tomography (SD-OCT), adverse events and number of injections administered.

ELIGIBILITY:
Inclusion Criteria:

* subfoveal or juxtafoveal CNV owing to AMD, defined by fluorescein angiography (FA)
* presence on SD-OCT of subretinal or intraretinal fluid associated or not with macular edema
* Best corrected visual acuity (BCVA) in the study eye between 20/20 and 20/125, inclusive
* total area of the lesion (including blood, neovascularization and scar/atrophy) of ≤8 disc areas, of which at least 50% must be active choroidal neovascularization (CNV) (defined as the neovascular component of the lesion as defined by FA
* all angiographic subtypes [predominantly classic, minimally classic and occult] were eligible)
* clear ocular media and adequate pupillary dilatation to allow collection of fundus photographs and FA of a sufficient quality to be analyzed
* intraocular pressure of 21 mmHg or less
* and no previous treatment for AMD

Exclusion Criteria:

* presence of scarring or atrophy >75% of the total lesion size (patients with subfoveal scar or atrophy were excluded)
* subretinal haemorrhage >75% of the total lesion size; presence of serous retinal pigment epithelial detachments >5 disc areas
* presence of intraocular inflammation (≥ trace cell or flare), epiretinal membrane, macular hole or vitreous haemorrhage
* history of idiopathic or autoimmune-associated uveitis in either eye
* significant media opacities, including cataract, which might interfere with VA, assessment of toxicity or fundus photography in the study eye
* presence of other causes of CNV, including pathological myopia (spherical equivalent of -3 diopters or more, or axial length of 25 mm or more, or fundus findings suggestive of pathologic myopia), ocular histoplasmosis syndrome, angioid streaks, choroidal rupture and multifocal choroiditis
* any retinal treatment (aside from antioxidants), including (but not limited to) intravitreal injections, photodynamic therapy with verteporfin, laser photocoagulation or surgery
* history of rhegmatogenous retinal detachment, pars plana vitrectomy or corneal transplant
* and previous radiation in the region of the study eye.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2010-11; Primary Completion 2012-03 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
mean VA change | 12 months
  change in ETDRS (early treatment diabetic retinopathy study) letters from baseline to 12 month-visit

SECONDARY OUTCOMES:
Percentage of patients with gain of ≥5, >10 and ≥15 letters ETDRS | 12 months
  percentage of patients with gain of ≥5, >10 and ≥15 letters ETDRS at 12 months compared to baseline
The percentage of patients losing <5, <15 and <30 ETDRS letters | 12 months
  percentage of patients with lost of <5, <15 and <30 ETDRS letters at 12 months compared to baseline
The mean VA | 6 and 12 months
  mean VA at 6 and 12 months in ETDRS letters
The median VA | 12 months
  median VA at 6 and 12 months in ETDRS letters
The mean number of injections | 12 months
  the mean number of injections administered to patients from baseline to month 12 ( month 12 not included)

CONTACTS AND LOCATIONS:
Overall Officials: Jordi M Mones, MD, Principal Investigator — Institut de la Macula i de la Retina
Locations (1):
- Institut de la Macula i de la Retina, Barcelona, Spain

REFERENCES:
- [Derived] Mones J, Biarnes M, Trindade F, Casaroli-Marano R. FUSION regimen: ranibizumab in treatment-naive patients with exudative age-related macular degeneration and relatively good baseline visual acuity. Graefes Arch Clin Exp Ophthalmol. 2012 Dec;250(12):1737-44. doi: 10.1007/s00417-012-2009-5. Epub 2012 Apr 15. PMID 22527314